CLINICAL TRIAL: NCT01877980
Title: Prediction of Uncuffed Endotracheal Tube Size in a Pediatric Population by Sonographic Measurements at Various Structures of the Airway Compared to Age-related Formulas and Little-finger Diameters
Brief Title: Ultrasound and Pediatric Endotracheal Tube Size
Acronym: SoTu2
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Christoph Schramm, M.D., Principal Investigator, Heidelberg University
Other Study IDs: S021/2013
Record Dates: First submitted 2013-06-05; First posted 2013-06-14 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Intubation With Uncuffed Endotracheal Tube

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study was to evaluate the ultrasonographic airway measurement in pediatric patients to compare the correct size of an uncuffed endotracheal tube (ETT) with the minimal transverse airway diameter (MTAD) with tube size predicted by different age-related formulas and diameter of little finger.

Previous studies already showed that a prediction of pediatric ETT is possible with the ultrasonographic measurement of the MTAD. In this study measurements are performed at three predefined anatomic structures of the airway with each of These at two airway pressures.

The investigators hypothesize that one of the specific measurements predicts the fitting ETT size better than age-related formulas or diameter of little finger.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent by the legal guadian
* elective surgery requiring endotracheal intubation

Exclusion Criteria:

* missing informed consent
* allergy to ultrasound gel

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Minimal transverse airway Diameter (MTAD) | Between administration of muscle relaxant and intubation (3min)
  In this study measurements of MTAD are performed at three predefined anatomic structures of the airway with each of these at two airway pressures in the time frame between the administration of muscle relaxant and Intubation (average time available 3min).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany